CLINICAL TRIAL: NCT01989936
Title: A Multicenter, Double - Blind, Randomized, Placebo - Controlled Parallel Group Study of the Efficacy and Safety of Oral Eletriptan (40 and 80mg) Given for the Treatment of Acute Migraine in Subjects Discontinued From Oral Sumatriptan
Brief Title: Eletriptan for the Treatment of Migraine in Patients With Previous Poor Response or Tolerance to Oral Sumatriptan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1601006
Record Dates: First submitted 2013-10-30; First posted 2013-11-21 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Migraine With or Without Aura
MeSH Terms: interventions — eletriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan 40 mg (Experimental)
  Interventions: Drug: Eletriptan 40 mg
- Eletriptan 80 mg (Experimental)
  Interventions: Drug: Eletriptan 80 mg

INTERVENTIONS:
Drug: Placebo — Subjects were randomized to one of the 3 treatment groups (eletriptan 40 mg, eletriptan 80 mg, or placebo) in a 2:2:1 ratio and were given sufficient medication to treat 3 migraine attacks (including a second dose for each attack for recurrence) within 18 weeks of the initial visit. Subjects were instructed to treat a moderate to severe migraine within 6 hours of the onset of pain provided the headache was not decreasing in severity, the aura phase had ended and they had taken no analgesic or antiemetic within 6 hours. Efficacy data was collected in a diary. Subjects were allowed to take rescue medication if they had no response to the study medication within 4 hours of onset.
  Arms: Placebo
Drug: Eletriptan 40 mg — Subjects were randomized to one of the 3 treatment groups (eletriptan 40 mg, eletriptan 80 mg, or placebo) in a 2:2:1 ratio and were given sufficient medication to treat 3 migraine attacks (including a second dose for each attack for recurrence) within 18 weeks of the initial visit. Subjects were instructed to treat a moderate to severe migraine within 6 hours of the onset of pain provided the headache was not decreasing in severity, the aura phase had ended and they had taken no analgesic or antiemetic within 6 hours. Efficacy data was collected in a diary. Subjects were allowed to take rescue medication if they had no response to the study medication within 4 hours of onset.
  Arms: Eletriptan 40 mg
Drug: Eletriptan 80 mg — Subjects were randomized to one of the 3 treatment groups (eletriptan 40 mg, eletriptan 80 mg, or placebo) in a 2:2:1 ratio and were given sufficient medication to treat 3 migraine attacks (including a second dose for each attack for recurrence) within 18 weeks of the initial visit. Subjects were instructed to treat a moderate to severe migraine within 6 hours of the onset of pain provided the headache was not decreasing in severity, the aura phase had ended and they had taken no analgesic or antiemetic within 6 hours. Efficacy data was collected in a diary. Subjects were allowed to take rescue medication if they had no response to the study medication within 4 hours of onset.
  Arms: Eletriptan 80 mg

SUMMARY:
To determine the tolerability and efficacy of eletriptan in patients who had discontinued oral sumatriptan due to lack of efficacy or intolerable adverse events (AEs) during previous clinical treatment (not a controlled trial).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age ≥ 18 years who met the International Headache Society (IHS) diagnostic criteria for migraine, with or without aura, and could reasonably expect to suffer at least one acute attack of migraine every 6 weeks.
* Subjects required to have discontinued therapy with oral sumatriptan at least 2 weeks, but not longer than 2 years, prior to the screening visit.
* Female subjects required to be adequately protected against pregnancy.

Exclusion Criteria:

* pregnancy or breastfeeding, known coronary artery disease, significant arrhythmias, heart failure, significant ECG abnormalities, and uncontrolled hypertension.
* Any significant systemic, organ, neurological, endocrine, metabolic, and psychological disorders reported by the patient or discovered during the physical examination
* Subjects considered to have atypical migraine such as frequent attacks, prolonged aura or any migraine that was considered atypical.
* Subjects who, during the course of the trial, required treatment with sumatriptan or any other 5-HT1B/1D agonist in addition to study medication.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 1999-01; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was 2-h headache response after taking the first dose of study medication for the first attack | 18 weeks
  Subjects recorded the intensity of each migraine headache in the diary based on a 4-point scale: 0, pain absent; 1, mild pain; 2, moderate pain; 3, severe pain. A response was considered a change from severe or moderate pain to mild or absent at various time points after dosing with study medication

SECONDARY OUTCOMES:
Sustained response was defined as achieving a headache response within 2 h post dose, with no recurrence or rescue medication needed | 18 weeks
  Recurrence was defined as a return of headache to moderate or severe intensity within 2-24 h if the subject had an initial response within 2 h of taking the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- Denmark (8):
  - Arhus Kommunehospital, Arhus C
  - Bispebjerg Hospital, Copenhagen
  - Centralsygehuset I Esbjerg, Esbjerg
  - Kas Glostrup, Glostrup Municipality
  - Hilleroed Sygehus, Hilleroed
  - Knud Kjaersgaard Pedersen, Hjørring
  - Neubauer, Ole (Private Practice), Nykoebing F
  - Korsgaard, Anne G. (Private Practice), Odense C
- Finland (7):
  - Haukiputaan Laakarikeskus, Haukipudas
  - Helsinki University Central Hospital, Helsinki
  - Hyvinkaa District Hospital, Hyvinkää
  - Torikeskuksen Laakariasema, Jyväskylä
  - Mikkelin Paansarkypoliklinikka (Mikkeli Headache), Mikkeli
  - Porin Laakarikeskus, Pori
  - Turku Headache Centre, Turku
- Netherlands (2):
  - Bosch Medicentrum (Locatie Willem Alexander Ziekenhuis), 's-Hertogenbosch
  - Sint Lucas Andreas Ziekenhuis (Location: St.Lucas), Amsterdam
- Norway (4):
  - Sentralsykehuset I Akershus, Nordbyhagen
  - Private Practice, Oyvind Rosjo, Oslo
  - Volvat Medisinske Senter, Oslo
  - Strandquist, Dr. Stein Bror, Tønsberg
- Sweden (7):
  - Migranklinik-Goeteborg, Gothenburg
  - Neurologsektionen, Lasarettet, Helsingborg
  - Neuro Kliniken, Helsingborg, Helsingborg
  - Medicin Kliniken, Sjukhuset, Kristinehamn
  - Medicin Kliniken, Universitetssjukhuset, Lund
  - St Gorans Sjukhus, Stockholm
  - Kronobergskliniken, Vaxjo
- Country not given (15):
  - Danderydssjukhus
  - Foretagshalsovarden Linden
  - Fylkessjukehuset I Molde
  - Huslakargruppen
  - Lakarhuset Hermelinen
  - Lakarhuset
  - Limhamns Lakargrupp, Tarnan
  - Lundsbysjukhus
  - Medicinskt Centrum
  - Nijmeegs Interkonfessioneel Ziekenhuis Canisius-Wilhelmina
  - Primarvarden
  - Regionsykehuset I Trondheim
  - Sentralsjukehuset I Hedmark
  - Sint Anna Ziekenhuis
  - Vardcentralen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601006&StudyName=Eletriptan%20for%20the%20Treatment%20of%20Migraine%20in%20Patients%20with%20Previous%0APoor%20Response%20or%20Tolerance%20to%20Oral%20Sumatriptan